CLINICAL TRIAL: NCT01463332
Title: Effect of Dexmedetomidine on Pain Due to Propofol Injection:A Randomised, Double-blind, Controlled Clinical Trial
Brief Title: Effect of Dexmedetomidine on Pain Due to Propofol Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KVG Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Shivakumar M C, MD, Assistant Professor, KVG Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMC/CT/3/2011; KVGMCH/CT/2/2011 (Other: KVG Medical college and hospital)
Record Dates: First submitted 2011-09-30; First posted 2011-11-01 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Pain; Intravenous Propofol Injection
Keywords: Propofol; Pain; Dexmedetomidine
MeSH Terms: conditions — Pain | interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group NS (Placebo Comparator): Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group NS were injected intravenously with 10 ml of normal saline before injection of propofol.
  Interventions: Drug: I.V injection of 10 ml normal saline
- Group D25 (Active Comparator): Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group D25 were injected intravenously with 0.25mic/kg of dexmedetomidine diluted with normal saline into 10ml before injection of propofol.
  Interventions: Drug: I.V injection with 0.25mic/kg of dexmedetomidine
- Group D50 (Active Comparator): Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group D50 were injected intravenously with 0.50mic/kg of dexmedetomidine diluted with normal saline into 10ml before injection of propofol.
  Interventions: Drug: I.V injection of 0.50mic/kg of dexmedetomidine

INTERVENTIONS:
Drug: I.V injection of 10 ml normal saline — Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group NS were injected intravenously with 10 ml of normal saline before injection of propofol.
  Other Names: Group NS
  Arms: Group NS
Drug: I.V injection with 0.25mic/kg of dexmedetomidine — Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group D25 were injected intravenously with 0.25mic/kg of dexmedetomidine diluted with normal saline into 10ml before injection of propofol.
  Other Names: dexmedetomidine
  Arms: Group D25
Drug: I.V injection of 0.50mic/kg of dexmedetomidine — Patients were randomly assigned in to three groups of 50 each using a computer-generated table of random numbers. Patients Group D50 were injected intravenously with 0.50mic/kg of dexmedetomidine diluted with normal saline into 10ml before injection of propofol.
  Other Names: Dexmedetomidine
  Arms: Group D50

SUMMARY:
Propofol is commonly used IV anesthetic, it has been formulated in a concentration of 10 mg/ml in a fat emulsion consisting of 10% soybean oil (long-chain triglycerides). When used for anesthetic induction, propofol causes pain on injection in 28%-90% of patients. pain probably results from a direct irritant effect. Several methods have been used to reduce this pain. Lidocaine pretreatment has been commonly proposed to decrease propofol induced pain, but its failure rate is between 13-32%. Dexmedetomidine is highly selective alfa-2 adrenoreceptor agonist. Alpha-2 receptors are located on blood vessels where they inhibit norepinephrine release. Investigators, therefore, speculated that dexmedetomidine could attenuate the pain due to injection of propofol. Investigators conducted a study to determine the efficacy of dexmedetomidine in decreasing pain due to injection of propofol.

DETAILED DESCRIPTION:
Propofol solution is fat emulsion consisting of soyabean oil. When used for anesthetic induction, propofol causes pain or discomfort on injection. Many factors appear to affect the incidence of pain, which includes site of injection, size of vein, speed of injection, buffering effect of blood, temperature and composition of propofol solution and concomitant use of drugs such as local anaesthetics and opiates.

Pain on injection of propofol can be immediate or delayed. Immediate pain probably results from a direct irritant effect whereas delayed pain probably results from an indirect effect via the kinin cascade. Delayed pain has latency of between 10 and 20 s. The pain produced is usually described as tingling, cold, or numbing, at its worst, a severe burning pain proximal to the site of injection. This sensation tends to occur within 10-20 s of injection and lasts only for the duration of injection. Despite this discomfort, the incidence of phlebitis is less than 1%.

Several methods have been used to reduce this pain with limited success. Lidocaine pretreatment is commonly used to decrease propofol induced pain, but its failure rate is between 13-32%.

Dexmedetomidine is an selective alfa-2 adrenoreceptor agonist with supraspinal, spinal, and peripheral actions. Alpha-2 receptors are located on blood vessels where they inhibit norepinephrine release. Investigators, therefore, speculated that dexmedetomidine could attenuate the pain due to injection of propofol.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* Both gender
* Age 18-60
* Elective surgery

Exclusion Criteria:

* Patients taking sedatives or analgesics in the past 24 hours
* History of allergic reactions to anesthetic drugs,
* Atrio-ventricular conduction defects
* Cardiovascular disease and
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Pain score after propofol injection | upto 24 hours
  After injecting study drugs the pain score after propofol was assessed by using visual rating scale and given score according to severity of pain 0 = no pain,
  1. = mild pain or soreness,
  2. = moderate pain and
  3. = severe pain associated with facial grimacing, arm withdrawal, movement or both.

SECONDARY OUTCOMES:
Incidence of Pain recall in postoperative recovery room | Upto 24 hrs.
  All patient were observed for 2-hrs in recovery room and were asked to recall if there was pain during injection of propofol in the recovery room and incidence of pain was graded as
  0-No recall of pain
  1-Recall of pain present.

CONTACTS AND LOCATIONS:
Overall Officials: Shivakumar M C, MD, Principal Investigator — KVG Medical College and Hospital